CLINICAL TRIAL: NCT00750204
Title: Airway Pressure Release Ventilation in Acute Lung Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NA_00017371
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome; Mechanical Ventilation
Keywords: Acute Lung Injury; ALI; Acute Respiratory Distress Syndrome; Mechanical Ventilation; Sedation; Critical Illness; Ventilator Induced Lung Injury; VILI; Cytokines; Protective Ventilation; Airway Pressure Release Ventilation; APRV; Breathing Comfort; Dyssynchrony; Asynchrony
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Critical Illness; Ventilator-Induced Lung Injury | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APRV (Experimental): Patients will be randomized to either arm. After 24 hours they will crossover to the alternative arm of the study for an additional 24 hours. After a total of 48 hours (24 hours in each study arm) the study will conclude.
  Interventions: Device: APRV
- Conventional MV (Active Comparator): Patients will be randomized to either arm. After 24 hours they will crossover to the alternative arm of the study for an additional 24 hours. After a total of 48 hours (24 hours in each study arm) the study will conclude.
  Interventions: Device: Conventional MV

INTERVENTIONS:
Device: APRV — APRV Protocol
  * Set fraction of inspired oxygen (FiO2) at 0.1 higher than the setting on conventional MV currently used
  * Tlow = 1.0 second (this setting shall remain unchanged throughout the trial).
  * Respiratory rate (RR) to equal 60-65% of RR on conventional MV.
  * P high = the inspiratory plateau pressure. Maximum P high = 30 cm H20.
  * Plow = 5 cm water (H2O). Adjust Plow to achieve pressure release volumes 5.5-6.5 ml/kg of percent body weight (PBW).
  * If release volumes on APRV are greater than desired, increase Plow by 2-4 cm H2O increments to a maximum of Plow = 12 cm H2O. If release volumes are larger than desired despite raising Plow to 12 cm H20, decrease P high in increments of 2-4 cm H20 to achieve desired release volumes (minimum P high = 12 cm H20). If release volumes on APRV still remain larger than desired,the participant will be excluded from the study and placed on conventional MV.
  Other Names: Lung-protective ventilation; Airway Pressure Release Ventilation
  Arms: APRV
Device: Conventional MV — Low tidal-volume mechanical ventilation
  Other Names: Lung protective ventilation; conventional mechanical ventilation
  Arms: Conventional MV

SUMMARY:
The purpose of this study is to compare airway pressure release ventilation (APRV) to conventional mechanical ventilation (MV) in patients with acute lung injury (ALI) to determine if APRV can reduce agitation, delirium, and requirements for sedative medications. We will also compare markers of inflammation in the blood and lung to determine if APRV reduces ventilator-induced lung injury (VILI), compared to conventional mechanical ventilation.

The proposed study is a randomized, crossover trial. We plan to enroll 40 patients with ALI and randomize to APRV or conventional MV for 24 hours. After this time the patients will be switched to the alternative mode of ventilation (MV or APRV) for another 24 hours. To assess breathing comfort, at the end of each 24-hour period we will measure the amounts of sedative and analgesic medications used. We will also measure the concentrations of markers of inflammation in the blood and lung as measures of VILI. Finally, throughout the study we will compare the adequacy of gas exchange with APRV compared to conventional MV.

DETAILED DESCRIPTION:
Acute respiratory failure is common in patients with acute lung injury. MV re-establishes adequate gas exchange; it allows time for administration of antibiotics, for the host's immune system to fight infections, and for natural healing. Approximately 60% of ALI patients survive to hospital discharge (1). However, conventional approaches to MV in ALI frequently cause dyssynchrony between a patient's spontaneous respiratory efforts and the ventilator's respiratory cycle (2;3). Dyssynchrony causes discomfort, anxiety, and agitation. To manage dyssynchrony, physicians frequently prescribe large doses of sedative and analgesic medications. These medications contribute to delirium and sleep deprivation during the critical illness, and may delay weaning from MV and discharge from the intensive care unit (2;4). They may also contribute significantly to neuromuscular and neurocognitive sequelae after recovery from ALI (5;6). Moreover, MV may itself cause additional lung injury (ventilator-induced lung injury, VILI) which could, paradoxically, delay or prevent recovery from respiratory failure in some ALI patients (7;9).

Airway pressure release ventilation (APRV) is a mode of MV that is designed to reduce patient-ventilator dyssynchrony and VILI. It differs from most other modes of MV in that it allows patients to breathe spontaneously at any time, independent of the ventilator's cycle. This feature may improve breathing comfort by minimizing patient-ventilator dyssynchrony. Improving comfort and reducing agitation may ultimately curtail the use of sedative and analgesic medications. Since a substantial proportion of ventilation results from the patient's spontaneous efforts independent of the ventilator cycle, the frequency of mechanically assisted breaths can be reduced. This may reduce VILI from the cyclic opening-closing of alveoli and small bronchioles that results from assisted MV breaths. Another feature of APRV that distinguishes it from other modes of MV is that it applies a sustained high pressure during inspiration and a brief period of lower pressure during exhalation. This approach may maximize and maintain alveolar recruitment throughout the ventilatory cycle while limiting high airway pressures, thus further reducing VILI. Moreover, spontaneous contractions of the diaphragm during APRV may open dependent atelectatic lung regions, improving ventilation-perfusion (V/Q) matching and gas exchange. However, these potential advantages of APRV are unproven.

ELIGIBILITY:
Inclusion Criteria:

Acute onset of:

1. Arterial Pressure of Oxygen (PaO2) / FiO2 ≤ 300
2. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph. The infiltrates may be patchy, diffuse, homogeneous, or asymmetric
3. Requirement for positive pressure ventilation via endotracheal tube, and
4. No clinical evidence of left atrial hypertension.
5. Receiving conventional MV, or lung-protective ventilation (LPV), in the assist control (AC) mode with positive end-expiratory pressure (PEEP) > 5 cm H2O Criteria 1-3 must occur within a 24-hour period. "Acute onset" is defined as follows: the duration of the hypoxemia criterion (#1) and the chest radiograph criterion (#2) must be < 7 days at the time of randomization.

Exclusion Criteria:

1. FiO2 > 70% or PaO2/FiO2 < 125 or arterial pH < 7.25
2. Greater than 6 days since all inclusion criteria are met
3. Anticipated to begin weaning from MV within 48 hours
4. Neuromuscular disease that prevents the ability to generate spontaneous tidal volumes.
5. Glasgow Coma Scale (GCS) < 15 within 1 week of intubation
6. Acute stroke (vascular occlusion or hemorrhage)
7. Current alcoholism or previous daily use of opioids or benzodiazepines before hospitalization
8. Acute meningitis or encephalitis
9. Pregnancy (negative pregnancy test required for women of child-bearing potential) or breast-feeding.
10. Severe chronic respiratory disease
11. Previous barotraumas during the current hospitalization
12. Clinical evidence of bronchoconstriction on bedside examination (i.e., wheezing).
13. Patient, surrogate, or physician not committed to full support
14. Severe chronic liver disease (Child-Pugh Score B or C)
15. International Normalized Ratio (INR) > 2.0
16. Platelet level < 50,000
17. Mean arterial pressure < 65, or patient receiving intravenous vasopressors (any dose of epinephrine, norepinephrine, phenylephrine, or dopamine > 5 mcg/kg/min)
18. Age < 16 years old
19. Morbid obesity (greater than 1kg/cm body weight).
20. No consent/inability to obtain consent
21. Unwillingness of the clinical team to use conventional low tidal-volume protocol for MV.
22. Moribund patient not expected to survive 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2008-10-15 (Actual); Study Completion 2008-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy G Brower, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital Medical Intensive Care Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] Sassoon CS, Foster GT. Patient-ventilator asynchrony. Curr Opin Crit Care. 2001 Feb;7(1):28-33. doi: 10.1097/00075198-200102000-00005. PMID 11373508
- [Background] Thille AW, Rodriguez P, Cabello B, Lellouche F, Brochard L. Patient-ventilator asynchrony during assisted mechanical ventilation. Intensive Care Med. 2006 Oct;32(10):1515-22. doi: 10.1007/s00134-006-0301-8. Epub 2006 Aug 1. PMID 16896854
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Hopkins RO, Weaver LK, Pope D, Orme JF, Bigler ED, Larson-LOHR V. Neuropsychological sequelae and impaired health status in survivors of severe acute respiratory distress syndrome. Am J Respir Crit Care Med. 1999 Jul;160(1):50-6. doi: 10.1164/ajrccm.160.1.9708059. PMID 10390379
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Ranieri VM, Suter PM, Tortorella C, De Tullio R, Dayer JM, Brienza A, Bruno F, Slutsky AS. Effect of mechanical ventilation on inflammatory mediators in patients with acute respiratory distress syndrome: a randomized controlled trial. JAMA. 1999 Jul 7;282(1):54-61. doi: 10.1001/jama.282.1.54. PMID 10404912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants were enrolled
Groups:
- Airway Pressure Release Ventilation (APRV) First: Patients will be randomized to either arm. After 24 hours they will crossover to the alternative arm of the study for additional 24 hours. After a total of 48 hours (24 hours in each study arm) the study will conclude Airway Pressure Release Ventilation •Set FiO2 at 0.1 higher than the setting on conventional MV currently used •Tlow = 1.0 second (this setting shall remain unchanged throughout the trial). •Respiratory rate (RR) to equal 60-65% of RR on conventional MV. •Phigh = the inspiratory plateau pressure. Maximum Phigh = 30 cm H20. •Plow = 5 cm H2O. Adjust Plow to achieve pressure release volumes 5.5-6.5 ml/kg of PBW. •If release volumes on APRV are greater than desired, increase Plow by 2-4 cm H2O increments to a maximum of Plow = 12 cm H2O. If release volumes are larger than desired despite raising Plow to 12 cm H20, decrease Phigh in increments of 2-4 cm H20 to achieve desired release volumes (min Phigh = 12 cm H20). If release volumes on APRV still remain larger than desire
- Conventional MV First: Patients will be randomized to either arm. After 24 hours they will crossover to the alternative arm of the study for an additional 24 hours. After a total of 48 hours (24 hours in each study arm) the study will conclude.
  Conventional MV: Low tidal-volume mechanical ventilation
Period: Overall Study
Arm/Group | Airway Pressure Release Ventilation (APRV) First | Conventional MV First
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — study halted prematurely | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- APRV: Patients will be randomized to either arm. After 24 hours they will crossover to the alternative arm of the study for an additional 24 hours. After a total of 48 hours (24 hours in each study arm) the study will conclude.
  APRV: APRV Protocol
  * Set FiO2 at 0.1 higher than the setting on conventional MV currently used
  * Tlow = 1.0 second (this setting shall remain unchanged throughout the trial).
  * Respiratory rate (RR) to equal 60-65% of RR on conventional MV.
  * Phigh = the inspiratory plateau pressure. Maximum Phigh = 30 cm H20.
  * Plow = 5 cm H2O. Adjust Plow to achieve pressure release volumes 5.5-6.5 ml/kg of PBW.
  * If release volumes on APRV are greater than desired, increase Plow by 2-4 cm H2O increments to a maximum of Plow = 12 cm H2O. If release volumes are larger than desired despite raising Plow to 12 cm H20, decrease Phigh in increments of 2-4 cm H20 to achieve desired release volumes (minimum Phigh = 12 cm H20). If release volumes on APRV still remain larger than desire
- Total: Total of all reporting groups
Arm/Group | APRV | Conventional MV | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Amount of Sedatives Used
Time Frame: 48 hours
Population: Data was not collected for this outcome measure, as the study was terminated prematurely.
Arm/Group | APRV | Conventional MV
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | APRV | Conventional MV
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes